CLINICAL TRIAL: NCT02146131
Title: Multicenter, Prospective, Randomized Trial of Bronchoscopy With Ultrathin Bronchoscope and Radial Endobronchial Ultrasound (R-EBUS) With Fluoroscopy Versus Standard Fiberoptic Bronchoscopy (FB) With Fluoroscopy for Biopsy of Pulmonary Lesions
Brief Title: Ultrathin Bronchoscope and Radial Endobronchial Ultrasound (R-EBUS) With Fluoroscopy Versus Standard Fiberoptic Bronchoscopy (FB) (P00029233 )
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Olympus (Industry); Johns Hopkins University (Other); Medstar Health Research Institute (Other); Mayo Clinic (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 00029233
Record Dates: First submitted 2014-05-20; First posted 2014-05-23 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Lesions; Pulmonary Nodules; Pulmonary Mass
Keywords: Peripheral pulmonary lesions; Solitary pulmonary lesions; Multiple pulmonary lesions
MeSH Terms: conditions — Multiple Pulmonary Nodules | interventions — Fluoroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard FB with fluoroscopy (Active Comparator): Administration of moderate or deep sedation, introduction of standard adult bronchoscope into the airway. Following application of topical anesthesia on vocal cord, trachea, bronchoscope is advanced distally under direct visualization. Localization of the lesion using fluoroscopy followed by the acquisition of pathologic and cytologic specimens using standard bronchial brush and standard transbronchial biopsy forceps. Evaluation of acquired samples for pathology. Performance of a portable chest X-ray to look for pneumothorax (PTX).
  Interventions: Device: Standard FB with fluoroscopy
- R-EBUS with ultrathin bronchoscope (Active Comparator): Administration of moderate or deep sedation, introduction of ultrathin bronchoscope into the airway. Following application of topical anesthesia on vocal cord, trachea, bronchoscope is advanced distally under direct visualization. Attempt to definitively locate the lesion with mechanical R-EBUS probe.
  Acquisition of pathologic and cytologic specimens using standard bronchial brush and standard transbronchial biopsy forceps. Performance of a portable chest X-ray to look for PTX.
  Interventions: Device: R-EBUS with ultrathin bronchoscope

INTERVENTIONS:
Device: Standard FB with fluoroscopy — Technique used, to go through the patient's airway, locate and obtain samples from pulmonary lesions
  Arms: Standard FB with fluoroscopy
Device: R-EBUS with ultrathin bronchoscope — Technique used to go through the patient's airway and using radial ultrasound, locate and obtain samples from pulmonary lesions
  Arms: R-EBUS with ultrathin bronchoscope

SUMMARY:
The purpose of this study is to compare the yield of two methods for obtaining a lung tissue sample: Procedure #1: standard fiberoptic bronchoscopy (FB) with fluoroscopy, and Procedure #2: ultrathin bronchoscope procedure with fluoroscopy and radial endobronchial ultrasound (R-EBUS). These two procedures are similar in that they both: (1) enable your doctor to look inside your lungs with a device called a bronchoscope, and (2) Use fluoroscopy, which is a technique that uses X-rays to see your lungs.

This will give the doctor an opportunity to use either of the bronchoscopy methods described above and compare the tests to see if R-EBUS provides better results than standard bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a solid lung lesion 2-5cm identified on chest CT with the intention to undergo bronchoscopic evaluation. If the lesion is partially solid (ie there is a ground glass component) then the solid portion must make up >75% of the lesion and measure at 2-5cm.The decision to pursue biopsy will be made by the treating physician and agreed upon by the patient. This will include patients determined to have an intermediate risk of malignancy (5-65%) and those non-surgical candidate with higher risk lesions in need of diagnosis for alternative treatment. OR
2. Patients with a solid lung lesion 2-5cm identified on chest CT that are surgical candidates with a high probability of cancer (>65%) will be referred for surgical evaluation. If the lesion is partially solid (ie there is a ground glass component) then the solid portion must make up >75% of the lesion and measure at 2-5cm. If the patient refuses surgery or if the surgeon requests a definitive diagnosis prior to surgery the patient will have the option to be included in this study. All sites will use the same online calculator to document probability of malignancy.
3. Are at least 22 years old,
4. Lack Bleeding disorders, and
5. Are able to provide informed consent

Exclusion Criteria:

1. Patients with a pure ground-glass opacity identified on chest CT
2. Patients with endobronchial involvement seen on chest CT.
3. Patients who refuse to participate,
4. Are less than 22 years of age,
5. Lack fitness to undergo flexible bronchoscopy as determined by the bronchoscopist prior to procedure, and
6. Are unable to provide informed consent
7. Pregnant

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2014-07; Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nichole T Tanner, MD, M.S.C.R, Principal Investigator — Medical University of South Carolina
Locations (5):
- United States (5):
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University Saint Louis, St Louis, Missouri
  - Medical University of South Carolina, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- R-EBUS With Ultrathin Bronchoscope: Administration of moderate or deep sedation, introduction of ultrathin bronchoscope into the airway. Following application of topical anesthesia on vocal cord, trachea, bronchoscope is advanced distally under direct visualization. Attempt to definitively locate the lesion with mechanical R-EBUS probe.
  Acquisition of pathologic and cytologic specimens using standard bronchial brush and standard transbronchial biopsy forceps. Performance of a portable chest X-ray to look for PTX.
  R-EBUS with ultrathin bronchoscope: Technique used to go through the patient's airway and using radial ultrasound, locate and obtain samples from pulmonary lesions
Period: Overall Study
Arm/Group | Standard FB With Fluoroscopy | R-EBUS With Ultrathin Bronchoscope
Started | 170 | 169
Completed | 109 | 113
Not Completed | 61 | 56
Not completed — Physician Decision | 61 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard FB With Fluoroscopy | R-EBUS With Ultrathin Bronchoscope | Total
Number analyzed (Participants) | 109 | 113 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (11.2) | 70.1 (9.9) | 68.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 51 | 107
  Male | 53 | 62 | 115
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 26 | 55
  White | 76 | 85 | 161
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Yield of Procedures; Number of Positive Diagnosis of Pulmonary Lesions
Description: Diagnostic yield of standard FB with fluoroscopy using standard adult bronchoscope versus bronchoscopy using ultrathin bronchoscope in combination with R-EBUS with or without Guidesheath for lung lesions 2-5 cm.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
Measure: Number; unit: participants
Arm/Group | Standard FB With Fluoroscopy | R-EBUS With Ultrathin Bronchoscope
Number analyzed (Participants) | 109 | 113
participants
  Diagnostic | 51 | 62
  Non-Diagnostic | 58 | 51

ADVERSE EVENTS:
Time Frame: 3 years
Description: It does not differ.
Arm/Group | Standard FB With Fluoroscopy | R-EBUS With Ultrathin Bronchoscope
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/113
Other Adverse Events (participants affected / at risk) | 6/109 | 5/113
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard FB With Fluoroscopy (N=109) | R-EBUS With Ultrathin Bronchoscope (N=113)
Adverse Event (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5) — Patient diagnosed with a pneumothorax orexcessive bleeding as a result of a standard of care bronchoscopy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT02146131/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT02146131/ICF_001.pdf